CLINICAL TRIAL: NCT05378737
Title: A Multicenter, Open Phase I Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Characteristics of BAT8006 for Injection in Patients With Advanced Solid Tumors
Brief Title: Evaluate the Safety, Tolerability and Pharmacokinetic Characteristics of BAT8006 for Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BAT-8006-001-CR
Record Dates: First submitted 2022-04-17; First posted 2022-05-18 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- A/1.2mg/kg (Experimental): Drug：BAT8006 for Injection, 1.2mg/kg, Q3W（Dose escalation study）
  Interventions: Drug: BAT8006 for Injection
- B/2.4mg/kg (Experimental): Drug：BAT8006 for Injection, 2.4mg/kg, Q3W（Dose escalation study）
  Interventions: Drug: BAT8006 for Injection
- C/ 3.0mg/kg (Experimental): Drug：BAT8006 for Injection, 3.0mg/kg, Q3W（Dose escalation study）
  Interventions: Drug: BAT8006 for Injection
- D/ 3.6mg/kg (Experimental): Drug：BAT8006 for Injection, 3.6mg/kg, Q3W（Dose escalation study）
  Interventions: Drug: BAT8006 for Injection
- 93mg/m^2 or 84mg/m^2 (Experimental): Drug：BAT8006 for Injection, 93mg/m^2 or 84mg/m^2, Q3W（Dose extension study）
  Interventions: Drug: BAT8006 for Injection

INTERVENTIONS:
Drug: BAT8006 for Injection — Intravenous infusion, once every 3 weeks (Q3W), the recommended infusion time of the first cycle is ≥90 minutes, if no infusion reaction occurs, the subsequent cycle can be completed within 30~120 minutes.
  Other Names: Exatecan conjugate of recombinant humanized monoclonal antibody against folate receptor α for injection

SUMMARY:
Objectives: To evaluate the safety and tolerability of BAT8006 for injection in patients with advanced solid tumors, explore the maximum tolerated dose (MTD), and provide the recommended dose for subsequent clinical trials.

DETAILED DESCRIPTION:
In this multi-center, open, dose-increasing, dose-expanding Phase I clinical study, rapid titration and a "3+3" dose-increasing design were used to explore the safety, tolerability and PK characteristics of BAT8006 for injection in patients with advanced solid tumors. During the dose-escalation test, appropriate doses were selected for the extended study according to the previous study data.

ELIGIBILITY:
Inclusion Criteria:

* The following items were satisfied to be included in the study:

  1. Age 18 to 75 years old (including the boundary value), gender is not limited;
  2. Voluntarily sign informed consent;
  3. For different cohorts, subjects should meet the following requirements:

     3-1) Dose escalation studies: Patients must be histologically or cytologically confirmed, patients with advanced or metastatic solid tumors who have failed or have no effective standard therapy, and patients who are intolerant to or refuse standard therapy, given the different tumor species, as determined by the clinician; 3-2) Dose Extension Study: Cohort 1) Ovarian Cancer: (1) Patients with advanced or metastatic epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer diagnosed histologically or cytologically with no more than three lines of previous treatment; (2) platinum-resistant recurrent ovarian cancer as defined by the U.S. Gynecologic Oncology Group (GOG) criteria (disease progression or recurrence confirmed by imaging within 6 months after receiving platinum-containing chemotherapy). ③ The expression of FRα in tumor tissue was positive; Cohort 2) Other advanced solid tumors: (1) Patients with advanced or metastatic solid tumors confirmed histologically or cytologically, failed or intolerant to standard therapy, were included only in endometrial cancer, breast cancer, and non-small cell lung cancer. ② It can provide tumor tissues to detect FRα expression level; Cohort 3) Ovarian Cancer: Patients with histologically or cytologically confirmed platinum-resistant advanced or metastatic epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer with four or five previous lines of treatment, platinum-resistant recurrent ovarian cancer as defined by the U.S. Gynecologic Oncology Group (GOG) (imaging confirmation of disease progression or recurrence within 6 months after receiving platinum-containing chemotherapy). ③ The expression of FRα in tumor tissue was positive.
  4. At least one measurable tumor lesion is present according to RECIST1.1 criteria;
  5. The United States Eastern Cancer Consortium (ECOG) requires a score of 0 or 1;
  6. Expected survival assessed by investigators ≥12 weeks;
  7. Have adequate organ and bone marrow reserve function,
  8. Fertile female patients must have a negative serological pregnancy test within 7 days prior to the first dosing and be willing to use an effective birth control/contraceptive method to prevent pregnancy during the study period up to 6 months after the last dosing of the study. Male patients must consent to an effective contraceptive method during the study period and up to 6 months after the last dosing in the study; Postmenopausal women must have amenorrhea for at least 12 months before they are considered infertile;
  9. Dose escalation study: Willing to provide previously archived or fresh tumor tissue samples (if no tumor tissue has been archived in the past, and the researcher assays that there is a great risk for patients to retake primary or metastatic tumor tissue samples); Dose expansion studies: Be willing to provide previously archived or fresh tumor tissue samples that can be used to detect FRα expression levels;
  10. Able to understand the test requirements, willing and able to follow the test and follow-up procedures.

Exclusion Criteria:

* If you meet any of the following conditions, you will not be allowed to enter this test:

  1. Have received experimental drug therapy or participated in a clinical study of a medical device within 4 weeks before the first administration of the investigational drug;
  2. Received chemotherapy, radiotherapy, small molecule targeted therapy, biotherapy, endocrine therapy, immunotherapy and other anti-tumor therapy within 4 weeks before the first use of the investigational drug (if the drug's 5x half-life is less than 28 days, the investigator and sponsor may decide whether to include the drug based on its pharmacological characteristics after discussion), except for the following: ① nitrosourea or mitomycin C within 6 weeks before the first use of the study drug; Oral fluorouracil is taken within 2 weeks prior to the first use of the study drug or within 5 half-lives of the drug (whichever is longer); (3) Chinese medicine/proprietary Chinese medicine with clear anti-tumor effects, immunomodulatory drugs (including but not limited to thymosin, interferon, interleukin, etc.) were systematically treated within 2 weeks before the first use of the investigational drug; (4) Palliative radiotherapy was performed within 2 weeks before the first use of the investigational drug;
  3. Grade ≥3 AE (graded using CTCAE v5.0) that were drug-related or of unknown relevance after prior treatment with any topoisomerase I inhibitor, such as irinotecan;
  4. Before the first administration of the investigational drug, AE (CTCAE5.0) from previous antitumor therapy still had grade 1, except in the following cases: a. Hair loss; b Pigmentation; c. Patients with distal toxicity caused by chemotherapy and radiotherapy who can not be further recovered by judgment; d. stable hypothyroidism with hormone replacement therapy;
  5. Patients who had undergone major surgery or had not recovered from surgery within 4 weeks prior to the first administration of the study drug, or had significant trauma, or required elective surgery during the trial period;
  6. Patients with a history of allogeneic cell or solid organ transplantation;
  7. Patients with primary central nervous system tumors or symptomatic central nervous system metastases, meningeal metastases or a history of epilepsy. Patients with asymptomatic or asymptomatic central nervous system metastases under clinical control or who have symptoms but are judged to be stable by the investigators can be included, provided that the following conditions are met :a. The clinical symptoms were stable ≥4 weeks before the first dose. b. Brain MRI enhancement showed no evidence of progression of central nervous system disease within 4 weeks prior to initial administration; c. Antiepileptic drugs have been stopped ≥2 weeks before the first administration, prednisone dosage ≤10mg/ day or equivalent dose of hormone;
  8. Other active malignancies within 5 years prior to first administration. Except locally cured tumors (e.g. basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer or carcinoma in situ of the breast, etc.);
  9. The following cardiovascular diseases occurred within 6 months before the first medication: New York Heart Association rating (NYHA) for symptomatic heart failure of grade 2 or higher, left ventricular ejection fraction (LVEF) < 50%, unstable arrhythmia or unstable angina, myocardial infarction requiring treatment, pulmonary embolism, uncontrolled hypertension (this protocol is defined as, despite the use of optimal antihypertensive therapy, However, systolic blood pressure > 160mmHg and/or diastolic blood pressure > 100mmHg after treatment were clinically significant as assessed by the investigator);
  10. Have any other medical condition, physical examination or laboratory results that, in the judgment of the investigator, are unsuitable for the use of the investigatory drug;
  11. Patients who have a history of non-infectious pneumonia/pulmonary inflammation requiring glucocorticoid therapy, or who currently have interstitial lung disease/pneumonia, or who cannot be ruled out by imaging during the screening period;
  12. Subjects requiring or being treated for tuberculosis, including but not limited to tuberculosis; Patients who have received standardized anti-tuberculosis treatment and have been confirmed cured by the researchers can be included;
  13. Severe infection within 4 weeks or active infection within 2 weeks prior to the first dose;
  14. The presence of persons infected with the following diseases: human immunodeficiency virus (HIV); Active hepatitis B virus infection [hepatitis B surface antigen (HBsAg) positive, HBV deoxyribonucleic acid (HBV-DNA) test >200 IU/ml or 103 copies /ml]; Hepatitis C virus infection [HCV antibody and viral ribonucleic acid (HCV-RNA) test positive]; Treponema pallidum antibody positive and RPR positive;
  15. Known hypersensitivity or delayed anaphylaxis to any of the components of the investigational drug;
  16. Those who are known to have experienced grade 3 or greater allergic reactions to macromolecular protein preparations/monoclonal antibodies;
  17. Patients with uncontrolled pleural effusion, pericardial effusion or abdominal effusion, or who require drainage;
  18. At risk of thrombosis or bleeding:

      1. A cerebrovascular accident or transient ischemic attack occurred within 6 months before the first dose;
      2. A history of deep vein thrombosis, pulmonary embolism, or any other severe thromboembolism within the 3 months prior to initial administration (implantable intravenous port or catheter-derived thrombosis, or superficial venous thrombosis is not considered "severe" thromboembolism);
      3. Any life-threatening bleeding event or grade 3 or 4 gastrointestinal/varicose bleeding event requiring blood transfusion, endoscopic or surgical treatment within 3 months prior to initial dosing;
      4. other diseases that the investigator believes have a higher risk of future bleeding or thrombosis;
  19. The presence of any other serious underlying medical condition (e.g., uncontrolled diabetes, active gastric ulcers, uncontrolled convulsive attacks, coagulopathy with severe signs or symptoms);
  20. A known history of mental illness, substance abuse, alcohol abuse or drug use that affected the results of the test;
  21. Women who are pregnant or breastfeeding or women or men who are preparing to give birth;
  22. The patient's compliance to participate in this clinical study is estimated to be insufficient or the investigator believes that there are other factors that are not suitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2025-12-08 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | At the end of Cycle 1 (each cycle is 21 days)
  DLT refers to any grade 3 or higher toxicities associated with the test drug that occurred within 21 days of the subject's initial administration
Maximum tolerated dose (MTD) | At the end of Cycle 1 (each cycle is 21 days)
  MTD was defined as exploration in a dose group observed ≤1/6 of subjects during the DLT evaluation period to the highest dose level of DLT.

SECONDARY OUTCOMES:
Pharmacokinetics（PK） | The first 6 treatment cycles(each cycle is 21 days)
  Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, Principal Investigator — The First Hospital of Jilin University
Locations (17):
- China (17):
  - Anhui Cancer Hospital, Hefei, Anhui
  - Beijing Obstetrics and Gynecology Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-Sen Memorlal Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Cancer Hospital Chinese Academy of Medical Sciences, Shenzhen Center, Shenzhen, Guangdong
  - Guangxi Medical University Cancer Hospital & Guangxi Cancer Institute, Nanning, Guangxi
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College of Hust, Wuhan, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital&Institute, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality